CLINICAL TRIAL: NCT04247997
Title: Effect of Disconnecting Pulmonary Vagus Nerve Branch on Chronic Cough After Unilateral Thoracoscopic Lobectomy: a Single-center, Randomized ,Single-blind, Controlled Trial
Brief Title: Effect of Disconnecting Pulmonary Vagus Nerve Branch on Chronic Cough After Unilateral Thoracoscopic Lobectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Han Yuan (Other)
Responsible Party: Sponsor-Investigator, Han Yuan, Doctor-in-charge of Anesthetist, Xuzhou Medical University
Organization: Xuzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XYFY2019-KL179-01
Record Dates: First submitted 2019-11-27; First posted 2020-01-30 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Postoperative Chronic Cough
Keywords: postoperative chronic cough; pulmonary vagus nerve branch; autonomic nervous system; pulmonary nerves; thoracoscopic lobectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group D (Experimental): disconnect pulmonary vague nerve branches
  Interventions: Procedure: disconnect pulmonary vague nerve branches
- Group P (No Intervention): preserve the pulmonary vague nerve branches

INTERVENTIONS:
Procedure: disconnect pulmonary vague nerve branches — When the operation is in the right side, the Azygous vein bow is used as the marker, and in the left side, the aortic arch is used as the marker to identify the vagus nerve trunk.Then the surgeons dissect the vagus nerve trunk. This is used as a clue to find the vagus nerve pulmonary branch leading to the hilum. The position of the detachment is after the anterior and posterior pulmonary branches of the vagus nerve separating from the trunk and before the formation of the lung plexus.
  Arms: Group D

SUMMARY:
The purpose of this study was to determine whether disconnecting pulmonary vagus nerve branch can abatement chronic cough in patients undergoing unilateral thoracoscopic lobectomy,compared with preserving pulmonary vagus nerve branch.

DETAILED DESCRIPTION:
After screening for the Inclusion criteria and the exclusion criteria, 116 patients undergoing unilateral thoracoscopic lobectomy are randomly assigned to two groups, disconnecting pulmonary vague nerve branches and preserving pulmonary vague nerve branches. The incidence of chronic cough after surgery is compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with preoperative imaging of bronchial lung cancer below the secondary bronchus ,the maximum diameter of the tumor ≤ 5cm (T ≤ 2) and staging check not suggesting distant and mediastinal lymph node metastasis (N ≤ 1, M = 0) schedule to receive elective unilateral thoracoscopic lobectomy from 2019 to 2021 will be included in the trial.
* ASAⅠ-Ⅲ

Exclusion Criteria:

* Chronic cough (>8 weeks), its causes including chronic bronchitis, asthma, gastroesophageal reflux disease, history of postnasal drip syndrome, and the use of ACEI drugs and so on;
* other history of lung surgery;
* patients with severe arrhythmia;
* there are contraindications for anesthesia and surgery;
* pregnancy and lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
The incidence of chronic cough after surgery | 3 months after surgery
  More than 8 weeks after surgery, there is no clear cause of cough with stable chest CT excluding the diagnosis of postnasal drip syndrome, asthma or the use of Angiotensin-converting enzyme inhibitor(ACEI), etc.

SECONDARY OUTCOMES:
The incidence of chronic cough after surgery | 1 month after surgery
  More than 8 weeks after surgery, there is no clear cause of cough with stable chest CT excluding the diagnosis of postnasal drip syndrome, asthma or the use of Angiotensin-converting enzyme inhibitor(ACEI), etc.
The score of the LCQ-MC scale after surgery | 1 month and 3 months after surgery
  The LCQ-MC was designed for the assessment of a chronic cough, consists of 19 items and three domains.
Length of operation | during the operation
volume of bleeding | during the operation
volume of postoperative drainage | within 30 days after surgery
the frequence of perioperative arrhythmia | during the operation
the incidence of Postoperative complication | within 30 days after surgery
  pulmonary complications, intestinal obstruction, pulmonary embolism, acute respiratory failure, acute renal failure, wound infection, cerebrovascular accident
the score of Cough symptom | postoperative 1 day,2 days,3 days,4 days,5 days,6 days
  The score was used to record daily symptom score for cough severity.The scale is scored by 4 levels at day and night respectively.The higher score means worse symptom.
the time of extubation | within 30 days after surgery
the incidence of gastrointestinal symptoms | within 3 months after surgery
  gastrointestinal symptoms include anorexia, belching, reflux, diarrhea, nausea
the incidence of postoperative hospitalization | within 30 days after surgery
pulmonary function 30 months after surgery | 30 months after surgery
  maximal voluntary ventilation, diffusing capacity of the lungs for carbon monoxideand forced expiratory volume

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

REFERENCES:
- [Derived] Zhang Q, Ge Y, Sun T, Feng S, Zhang C, Hong T, Liu X, Han Y, Cao JL, Zhang H. Pulmonary vagus nerve transection for chronic cough after video-assisted lobectomy: a randomized controlled trial. Int J Surg. 2024 Mar 1;110(3):1556-1563. doi: 10.1097/JS9.0000000000001017. PMID 38116674